CLINICAL TRIAL: NCT06528509
Title: An Artificial-intelligence-powered Intervention to Aid the Informed Consent Process for Cataract Surgery for English Speaking and Bengali Speaking Patient Population Groups: A Mixed-methods Randomised Control Trial
Brief Title: AI-Enhanced Consent for Cataract Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Medical Protection Society Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KANS1002
Record Dates: First submitted 2024-07-05; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cataract
Keywords: Cataract surgery; Complaints; Litigation; Informed consent
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: The study is designed as a parallel, randomized controlled trial. Participants scheduled for cataract surgery are randomly allocated into two groups: the intervention group and the control group. The intervention group receives AI-generated informative videos, while the control group receives standard written information brochures. The study will run in two cohorts, with Cohort A including English speaking patients and Cohort B Bengali speakers.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care Providers: The clinicians responsible for confirming consent on the day of surgery will be blinded to the group assignments of the patients. They will not know whether a patient received the AI-generated video or the standard written information brochure.
  Outcomes Assessors: The individuals assessing the outcomes, including patient understanding and satisfaction, as well as preoperative anxiety levels, will also be blinded to the group assignments. This includes the personnel administering and analyzing the multiple-choice questionnaires and anxiety scales.
  Participants: Participants will not be blinded as they will be aware of the type of information they received (AI-generated video or written brochure).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Generated Informative Videos (Experimental): Participants in this arm will receive an AI-generated informative video. The video will provide comprehensive information about cataract surgery, including the procedure, risks, benefits, and postoperative care. The content will be generated using the Synthesia platform, which uses artificial intelligence to create realistic, photo-realistic digital avatars to deliver the information. The aim is to improve patient understanding, satisfaction, and reduce preoperative anxiety compared to traditional information delivery methods. The video will be produced in English for Cohort A, and translated into Bengali for Cohort B.
  Interventions: Behavioral: AI-Generated Informative Videos
- Standard Written Information Brochures (Active Comparator): Participants in this arm will receive the standard information provided to patients undergoing cataract surgery, which consists of written information brochures. These brochures include comprehensive details about the cataract surgery procedure, potential risks, benefits, and postoperative care. The brochures are designed to provide all necessary information to help patients make an informed decision regarding their surgery. The leaflet will be supplied in English for Cohort A, and Bengali for Cohort B.
  Interventions: Behavioral: Standard Written Information Brochures

INTERVENTIONS:
Behavioral: AI-Generated Informative Videos — Participants in the experimental arm will receive an AI-generated video designed to provide comprehensive information about cataract surgery. The video will cover key aspects of the procedure, including the nature of the surgery, potential risks, benefits, and postoperative care. The video will be produced in English for Cohort A, and translated into Bengali for Cohort B.
  The video will be delivered to participants via a secure link sent to their mobile devices or email. Patients can watch the video at their convenience, and they are encouraged to view it as many times as necessary to fully understand the information provided. The video link will be provided once after the initial clinic appointment, but patients can access and watch the video multiple times.
  The videos will be created using the Synthesia platform, which uses artificial intelligence to generate realistic, photo-realistic digital avatars that deliver the information in a personalized and engaging manner.
  Arms: AI-Generated Informative Videos
Behavioral: Standard Written Information Brochures — Participants in the control arm will receive traditional written information brochures about cataract surgery. These brochures are designed to deliver detailed and essential information in a clear and understandable format. The brochures will be handed to participants during their face-to-face clinic appointment. Patients can read the material at their convenience and keep it for future reference. These brochures follow standardized guidelines and recommendations to ensure that all relevant information is included and presented in an accessible manner. The leaflet will be supplied in English for Cohort A, and Bengali for Cohort B.
  Arms: Standard Written Information Brochures

SUMMARY:
This research focuses on enhancing the informed process for patients before undergoing cataract surgery. Currently, this process involves verbal discussions and written materials that may not fully address patients' understanding of the surgery, its risks, and benefits. This study aims to introduce an innovative approach using artificial intelligence (AI) to generate informative videos tailored to patients' needs, accounting for education level, ethnicity, and language barriers.

Why is this important? Informed consent is not just a legal requirement; but it's a fundamental patient right. Ensuring patients truly understand their treatment options leads to better satisfaction, both from the patient and clinician's perspective.

This study compares the effectiveness of AI-generated videos against traditional information delivery methods (information brochures). Patients scheduled for cataract surgery will experience either the new AI video approach or the standard process. The goal is to see if the videos lead to better understanding of the procedure and overall satisfaction. The investigators will be running the study in two parallel cohorts - with Cohort A involving an English speaking population, and Cohort B a Bengali speaking population with all patient facing materials translated into Bengali.

This research is crucial for patients seeking clarity about cataract surgery, for doctors aiming to improve patient care, and for researchers exploring patient education innovations. Funded by the Medical Protection Society (MPS), the investigators hope this intervention has broader effects such as reducing the number of complaints and litigations, improving the efficiency of consenting for surgery and delivering information, and improving theatre utilisation by reducing last minute cancellations.

DETAILED DESCRIPTION:
Background and Rationale

Cataract surgery is one of the most frequently performed procedures in the NHS, yet the process of obtaining informed consent remains a significant challenge. Traditional methods of informed consent, primarily involving verbal discussions and written materials, often fail to ensure that patients fully understand the surgery, its risks, and benefits. This is especially problematic for patients with limited health literacy, language barriers, or other socioeconomic factors that affect their ability to comprehend complex medical information.

Objectives

The primary objective of this study is to enhance the informed consent process for cataract surgery by using artificial intelligence (AI) to create personalized informative videos. These videos will be tailored to meet the specific needs of patients, taking into account their educational levels, language preferences, and cultural backgrounds. The AI-generated videos will be compared against traditional information delivery methods, such as verbal briefings and written brochures, to assess their effectiveness in improving patient understanding, satisfaction, and reducing anxiety.

Study Design

This study will be conducted with two cohorts, each targeting different patient demographics to assess the feasibility and effectiveness of the AI intervention.

Cohort A:

Focus on English-proficient patients. Participants will be randomized into two groups: one receiving the AI-generated video and the other receiving standard written brochures.

Cohort B:

Expand to a Bengali speaking population with limited English proficiency. Same randomized design as Cohort A.

Methods

Participants will be recruited from Moorfields Eye Hospital and will include 100 patients in each cohort. The study will use a mixed-methods approach, incorporating both quantitative and qualitative data collection.

Quantitative Measures:

A multiple-choice questionnaire will assess patient understanding of the surgery.

State Trait Anxiety Inventory (STAI) will measure patient anxiety levels. Time and motion studies will track the duration of information delivery and consent confirmation processes.

Cancellation rates and incidence of complaints or litigations will be recorded.

Qualitative Measures:

Semi-structured interviews will explore patient experiences with the information delivery methods, their engagement with digital tools, and their overall satisfaction with the consent process.

Anticipated Benefits:

* Improved patient understanding of cataract surgery, leading to higher satisfaction and reduced anxiety.
* Potential reduction in surgery cancellations and complaints, improving overall theatre utilization.
* Enhanced clinician satisfaction by streamlining the consent process and reducing the likelihood of malpractice claims.

Ethical Considerations:

The study will ensure that all AI-generated content is rigorously reviewed for accuracy and cultural sensitivity. Participants will be informed about the AI nature of the videos, and all data will be handled in compliance with GDPR regulations to ensure confidentiality and security. All materials in Cohort B will be checked by a native Bengali speaker with a medical background. The investigators will be using a validated Bengali translation of the State Trait Anxiety Inventory (STAI).

Dissemination Strategy

Findings from the study will be disseminated through various channels, including academic publications, presentations at national and international conferences, and reports to relevant healthcare authorities. The results will also be shared with participants and the broader public through social media and community engagement initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Have capacity to consent
* Listed for first time cataract surgery
* English speakers for Cohort A
* Bengali speakers for Cohort B

Exclusion Criteria:

* Previously undergone cataract surgery
* Partner who has undergone cataract surgery
* Below the age of 18
* Unable to utilise a device for watching information videos and completing quiz

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-11 (Estimated); Primary Completion 2025-09-11 (Estimated); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Information understanding and retention | One week after intervention
  Assessed via a 12-question multiple-choice quiz sent via text message one week after the initial appointment.

SECONDARY OUTCOMES:
Patient Anxiety Level | Baseline; pre-intervention
  Measured using the State Trait Anxiety Inventory (STAIT) at the initial consultation and on the day of surgery.
Patient Anxiety Level | On day of surgery
  Measured using the State Trait Anxiety Inventory (STAIT) at the initial consultation and on the day of surgery.
Time and Motion Study | On day of surgery
  Time taken for information delivery and consent confirmation on the day of surgery will be recorded.
Participant-reported engagement time with the information material | One week after intervention
  This will be added as a question following the information understanding and retention quiz.
Cancellation rates | Within 7 days of surgery
  Day-of surgery and short notice cancellation rates and reasons will be documented.
Incidence of incidents and complaints | Up to 12 months post-operatively
  Any complaints or formal claims related to the surgery will be followed up for 12 months post-operatively
Patient and clinician satisfaction: Assessed on the surgery day using a 5-point Likert scale Patient and clinician satisfaction | On day of surgery
  Assessed on the surgery day using a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Swan Kang, MBBS, MBioch (Oxon), FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Moorfields Eye Hospital Stratford, London
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers. This decision is based on concerns about participant privacy and confidentiality, as well as the sensitive nature of the data collected in this study such as patient anxiety levels, and complaints and litigations. Instead, we will disseminate aggregated findings through peer-reviewed publications and presentations, ensuring the protection of participant identities while sharing valuable insights with the scientific community.

REFERENCES:
- [Background] Ali N, Little BC. Causes of cataract surgery malpractice claims in England 1995-2008. Br J Ophthalmol. 2011 Apr;95(4):490-2. doi: 10.1136/bjo.2010.182774. Epub 2010 Aug 30. PMID 20805130
- [Background] Zhang Y, Ruan X, Tang H, Yang W, Xian Z, Lu M. Video-Assisted Informed Consent for Cataract Surgery: A Randomized Controlled Trial. J Ophthalmol. 2017;2017:9593631. doi: 10.1155/2017/9593631. Epub 2017 Jan 16. PMID 28191349
- [Background] Shukla AN, Daly MK, Legutko P. Informed consent for cataract surgery: patient understanding of verbal, written, and videotaped information. J Cataract Refract Surg. 2012 Jan;38(1):80-4. doi: 10.1016/j.jcrs.2011.07.030. Epub 2011 Nov 6. PMID 22062774
- [Background] Zhang MH, Haq ZU, Braithwaite EM, Simon NC, Riaz KM. A randomized, controlled trial of video supplementation on the cataract surgery informed consent process. Graefes Arch Clin Exp Ophthalmol. 2019 Aug;257(8):1719-1728. doi: 10.1007/s00417-019-04372-5. Epub 2019 May 30. PMID 31144057
- [Background] Wagner SK, Raja L, Cortina-Borja M, Huemer J, Struyven R, Keane PA, Balaskas K, Sim DA, Thomas PBM, Rahi JS, Solebo AL, Kang S. Determinants of non-attendance at face-to-face and telemedicine ophthalmic consultations. Br J Ophthalmol. 2024 Mar 20;108(4):625-632. doi: 10.1136/bjo-2022-322389. PMID 37217292
- [Background] Bhan A, Dave D, Vernon SA, Bhan K, Bhargava J, Goodwin H; Medical Defence Union; Medical Protection Society; Medical and Dental Defence Union of Scotland. Risk management strategies following analysis of cataract negligence claims. Eye (Lond). 2005 Mar;19(3):264-8. doi: 10.1038/sj.eye.6701493. PMID 15286671
- [Background] Mathew RG, Ferguson V, Hingorani M. Clinical negligence in ophthalmology: fifteen years of national health service litigation authority data. Ophthalmology. 2013 Apr;120(4):859-64. doi: 10.1016/j.ophtha.2012.01.009. Epub 2012 Mar 2. PMID 22386949
- [Background] Ali N. A decade of clinical negligence in ophthalmology. BMC Ophthalmol. 2007 Dec 20;7:20. doi: 10.1186/1471-2415-7-20. PMID 18096077
- [Background] Gill ZS, Caldwell AS, Patnaik JL, Marin AI, Mudie LI, Grove N, Ifantides C, Ertel MK, Puente MA, Seibold LK. Comparison of cataract surgery outcomes in English proficient and limited English proficiency patients. J Cataract Refract Surg. 2023 Jun 1;49(6):595-601. doi: 10.1097/j.jcrs.0000000000001164. PMID 36779806
- [Background] Patel DN, Wakeam E, Genoff M, Mujawar I, Ashley SW, Diamond LC. Preoperative consent for patients with limited English proficiency. J Surg Res. 2016 Feb;200(2):514-22. doi: 10.1016/j.jss.2015.09.033. Epub 2015 Oct 3. PMID 26541685